CLINICAL TRIAL: NCT01419002
Title: Neoadjuvant Radiotherapy in Patients With Primary Resectable Adenocarcinoma of the Pancreatic Head Plus Adjuvant Chemotherapy: a Randomized Controlled Phase III Trial
Brief Title: Study to Evaluate if Neoadjuvant Radiotherapy Improves Recurrence Free Survival in Pancreatic Head Cancer
Acronym: Net-Pac
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: lack of recruitment
Sponsor: CHIR-Net (Network)
Collaborators: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NetPac
Record Dates: First submitted 2011-08-13; First posted 2011-08-17 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: Pancreatic Cancer; Adenocarcinoma; Neoadjuvant Radiotherapy
MeSH Terms: conditions — Pancreatic Neoplasms; Adenocarcinoma | interventions — Surgical Procedures, Operative; Pancreaticoduodenectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neoadjuvant RTx (Experimental)
  Interventions: Radiation: neoadjuvant RTx
- Surgery (Active Comparator)
  Interventions: Procedure: Surgery

INTERVENTIONS:
Radiation: neoadjuvant RTx — Neoadjuvant radiotherapy with external intensity modulated beam radiation followed by duodenopancreatectomy and adjuvant chemotherapy according to German S3 guidelines.
  Other Names: Intensity modulated beam radiation (IMBR).
  Arms: Neoadjuvant RTx
Procedure: Surgery — Surgery and adjuvant chemotherapy according to German S3-guidelines
  Other Names: Kausch-Whipple, Pancreaticoduodenectomy, ppWhipple
  Arms: Surgery

SUMMARY:
Net-Pac investigates if radiation prior to surgical resection improves survival in patients with pancreatic head cancer without metastases.

DETAILED DESCRIPTION:
The trial is designed to show that neoadjuvant radiotherapy followed by surgery improves local recurrence free survival compared to surgery alone in patients with resectable adenocarcinoma of the pancreatic head.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the pancreatic head
* Age ≥ 18 years
* Signed informed consent
* ECOG performance status of 0-2

Exclusion Criteria:

* Curative resection is not feasible or presence of metastatic disease
* Patients not eligible for surgery (ASA ≥ 4)
* Participation in an other clinical trial
* Unable or unwilling to sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Local recurrence free survival | At 12 months postoperative

SECONDARY OUTCOMES:
Percentage of surgical R0-resections in both groups | Until 10 days postoperative
  Determined by histopathological analysis of the surgical specimen.
30-day morbidity and mortality | 30 day period after the operation
Toxicity of preoperative Radiotherapy | Start of the radiotherapy until 12 months postoperative.
  Number of patients with adverse events in both groups, number of adverse events in both groups and number of grade 3 and 4 adverse events according to the Common Terminology Criteria for Adverse Events version 3.0 (CTCAE v 3.0) in both groups
Clinical response rate (RECIST-criteria) and histological response rate | Until 1 year postOP
Time to tumor progression (local and systemic) | Until 1 year postoperative
Quality of life | Until 12 months postoperative
Overall survival after 1 year | Until 1 year postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Helmut M Friess, Prof. MD, Principal Investigator — Technical University of Munich; Michael Molls, Prof. MD, Study Director — Technical University of Munich
Locations (1):
- Klinikum rechts der Isar, Technische Universität München, Munich, Germany

REFERENCES:
- See also: Department of Radiation Oncology, Technische Universität München — http://tumstrahlen.einzelportal.de/